CLINICAL TRIAL: NCT03756038
Title: Single Dose Administration of Benzodiazepines to Reduce Distress, Pain Severity, and the Need for Opiates Both During and After Emergency Department Care
Brief Title: Benzodiazepines for the Reduction of Distress and Pain During and After Emergency Department Care
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: It was not feasible to enroll Emergency Department patients into this protocol
Sponsor: Maria Pacella (Other)
Collaborators: University of Pittsburgh Physicians (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Maria Pacella, Research Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO18090064
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Results first posted 2020-02-26 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Lorazepam

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to either the experimental condition (lorazepam) or the control condition (placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Drug: Oral Lorazepam (1mg) (Experimental): Lorazepam (Ativan) is indicated for the management of anxiety disorders or for the short-term relief of the symptoms of anxiety or anxiety associated with depressive symptoms.
  Interventions: Drug: Lorazepam
- Drug: Oral Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Placebos — In this study, patients will receive oral placebo, an inactive solution that looks like the study drug, but contains no active ingredients
  Arms: Drug: Oral Placebo
Drug: Lorazepam — The purpose of this study is to determine whether a single low dose of Lorazepam/Ativan (1mg) can relieve pain and reduce negative mood in the emergency department and for 2 weeks after emergency department treatment.
  Other Names: Ativan
  Arms: Drug: Oral Lorazepam (1mg)

SUMMARY:
In this proposal, the investigators will determine if a single dose of oral lorazepam reduces distress, pain severity, and need for opiate analgesics both in the ED and in the acute recovery period after discharge. The investigators will compare the lorazepam arm to a placebo arm.

DETAILED DESCRIPTION:
The investigators will enroll 120 medically stable adult patients who present to two emergency departments with a physical injury (< 24 hours ago) and a chief complaint of pain.

The investigators will randomly assign subjects using a blocked randomization schedule to either: 1) a single dose of oral lorazepam (1mg), or 2) oral placebo. Emergency department providers and patients will be blind to treatment allocation.

All participants will complete measures of negative affect and pain scores at baseline, and and 1 and 2 hours post-study drug administration. The investigators will record any analgesics administered in the emergency department until discharge. Patients will also undergo quantitative sensory testing in the Emergency Department at baseline, and after study drug administration. At 14-days post-discharge, the investigators will measure summary reports of pain, mood, and analgesic medication used.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18-65
* Sustained a physical injury with a pain score ≥ 5 on the numeric rating scale [NRS] from 0- 10 with anchors of 0 = "no pain" and 10 = "worst pain imaginable"
* Expected to be in the ED for at least 2 hours, in a private treatment room
* Ownership of a cell phone with text messaging capabilities
* Emergency Department admission assessment confirmed subject is not suicidal.

Exclusion Criteria:

* Non-English speaking
* Not medically suitable for lorazepam per treating MD (e.g. medical condition where benzodiazepines are contraindicated or may be unsafe)
* Not alert and oriented
* Active psychosis, self-injury, suicidal/homicidal intentions on initial evaluation by treating team
* Seeking treatment due to a mental health or substance use disorder
* History of chronic opioid use
* Prescribed opioid or benzodiazepine use within the past 24 hours
* Alcohol use within the past 12 hours or medical history of alcoholism.
* Clinical indication for open-label benzodiazepine administration in the ED.
* Any use of recreational narcotics throughout lifetime
* Sensitivity or allergy or intolerance to opioids or benzodiazepines
* Current neurological disease (e.g., multiple sclerosis, stroke, brain tumor, seizure disorder, etc.)
* Prisoner

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Pacella, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC Mercy Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided
here is no plan in place yet because it is undecided whether the research team will need to share the data with investigators/researchers not listed on the protocol.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug: Oral Lorazepam (1mg) | Drug: Oral Placebo
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to feasibility issues, we had to prematurely halt enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug: Oral Lorazepam (1mg) | Drug: Oral Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 48 [48 to 48] |  | 48 [48 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Severity in the Emergency Department: Numeric Rating Scale
Description: Pain Numeric Rating Scale (on a scale from 0, no pain to 10, worst pain imaginable)
Time Frame: The item is anchored to pain intensity "right now" at 60 minutes post-study drug administration
Population: No one was enrolled in the placebo group because we prematurely halted enrollment due to lack of feasibility
Measure: Number; unit: units on a scale
Arm/Group | Drug: Oral Lorazepam (1mg) | Drug: Oral Placebo
Number analyzed (Participants) | 1 | 0
units on a scale | 6 |

2. Secondary Outcome: Negative Affect in the Emergency Department
Description: Positive and Negative Affect Schedule (PANAS)-We will use the 10 items of the Negative Affect Scale; each of these items are scored on a Likert Scale ranging from 1 (very slightly/not at all) to 5 (extremely). The responses for each of the 10 items are summed to create the Negative Affect Score; scores may range from 10-50, with lower scores representing lower scores of negative affect.
Time Frame: The 10 items of the Negative Affect Scale are anchored to mood "right now" at 60 minutes post-study drug administration.
Population: No subjects were enrolled in the placebo group because enrollment was prematurely halted due to lack of feasibility
Measure: Number; unit: units on a scale
Arm/Group | Drug: Oral Lorazepam (1mg) | Drug: Oral Placebo
Number analyzed (Participants) | 1 | 0
units on a scale | 10 |

ADVERSE EVENTS:
Time Frame: 2-weeks of study duration
Description: There are 0 participants at risk in the placebo arm because no participants were enrolled to that arm.
Arm/Group | Drug: Oral Lorazepam (1mg) | Drug: Oral Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT03756038/Prot_SAP_000.pdf